CLINICAL TRIAL: NCT03494595
Title: Perioperative Thromboelastometry as a Predictor of Thrombotic Complications During Pediatric Recipient Liver Transplantation
Brief Title: Thromboelastometry as a Predictor of Thrombotic Complications During Pediatric Recipient Liver Transplantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hamada Hamed, Assistant Lecturer, Assiut University
Other Study IDs: TEG PLT
Record Dates: First submitted 2018-03-27; First posted 2018-04-11 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Pediatric Liver Transplantation
Keywords: Pediatric Liver Transplantation, Thromboelastometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Thrombosis: Patients who will develop thrombosis perioperatively
  Interventions: Procedure: Pediatric Liver transplantation
- No thrombosis: Patients who will not develop thrombosis perioperatively
  Interventions: Procedure: Pediatric Liver transplantation

INTERVENTIONS:
Procedure: Pediatric Liver transplantation — Pediatric Liver transplantation

SUMMARY:
The study aims to correlate the perioperative results of a device called thromboelastogram, which is used to detect coagulation abnormalities, with thrombotic complications during pediatric recipient liver transplantation.

DETAILED DESCRIPTION:
Pediatric patients undergoing liver transplant are at risk for significant bleeding and thrombotic complications. Studies in both pediatric and adult cohorts estimate an incidence of thrombotic events in up to 26% of cases. Hepatic artery and portal vein thrombosis (PVT) are reported at rates of 5-15% in pediatric cohorts, which is three to four times the incidence in adults. Bleeding estimates are harder to quantify given variability in the definition of major bleeding, but range from approximately 5 to 9%.The contribution of bleeding to morbidity is difficult to quantify, but thrombotic complications are known to reduce graft survival and contribute significantly to adverse outcomes, with mortality rates approaching 50% in those with hepatic artery thrombosis.

Thromboelastometry offers rapid, comprehensive, and global clinical assessment of the patients' coagulation status, as demonstrated by several studies.

Little data exists in the use of thromboelastography (TEG) in pediatric liver transplantation. In 2011, Curiel et al implemented pre-transplant TEGs for patients listed for liver transplantation. The invistigators sought to examine if there were any correlations with preoperative hypercoagulable indices on the TEG and postoperative thrombotic complications.The invistigators have identified that a preoperative hypercoagulable TEG portends to thrombotic complications in pediatric liver transplant patients. Further studies are needed to explore perioperative management strategies for high risk patients to prevent the development of postoperative thrombotic complications based upon preoperative TEG studies. That's why the invistigators will study the perioperative thromboelastometry as a predictor of thrombotic complications during pediatric recipient liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant must be between 3 months and 15 years of age.
* Participant is a recipient of a first liver allograft from living donors.
* Participant is a single-organ recipient (liver only).
* Participants' parent/guardian is capable of understanding the purposes and risks of the study and must sign an informed consent for the study.

Exclusion Criteria:

* Pre-existing blood disease.
* A history of liver transplantation.
* Multivisceral transplantation.
* Participants' parent/guardian refused to participate in the study.

Ages: 3 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatrics undergoing liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Intraoperative thrombotic events (hepatic artery or portal vein thrombosis) | Intraoperative, an average of 12 hours
  Any documented thrombus by imaging or clinical diagnosis made by direct observation during a surgical procedure. This includes both venous and arterial thromboembolic events.
Thrombotic events (hepatic artery or portal vein thrombosis) | Postoperative up to 1 week.
  Patients will be screened for hepatic thrombosis regularly with liver Doppler ultrasound during the first week postoperatively, with confirmatory imaging based on identified clinical or imaging concerns.

SECONDARY OUTCOMES:
Coagulation Time preoperative. | Preoperative up to 1 day before surgery.
  Coagulation Time (CT, in seconds), the time from the start of measurement until a clot firmness of 2 mm is detected by thromboelastometry preoperatively.
Coagulation Time in pre-anhepatic stage. | In pre-anhepatic stage, an average of 4 hours.
  Coagulation Time (CT, in seconds), the time from the start of measurement until a clot firmness of 2 mm is detected by thromboelastometry during pre-anhepatic stage.
Coagulation Time in anhepatic stage. | In anhepatic stage, an average of 2 hours.
  Coagulation Time (CT, in seconds), the time from the start of measurement until a clot firmness of 2 mm is detected by thromboelastometry during anhepatic stage.
Coagulation Time after reperfusion. | After reperfusion, an average of 4 hours.
  Coagulation Time (CT, in seconds), the time from the start of measurement until a clot firmness of 2 mm is detected by thromboelastometry after reperfusion.
Coagulation Time at the end of surgery. | At the end of surgery, an average of 12 hours.
  Coagulation Time (CT, in seconds), the time from the start of measurement until a clot firmness of 2 mm is detected by thromboelastometry at the end of surgery.
Clot Formation Time preoperative | Preoperative up to 1 day before surgery.
  Clot Formation Time (CFT, in seconds), the time needed to increase clot firmness from 2 to 20 mm amplitude as detected by thromboelastometry preoperatively.
Clot Formation Time in pre-anhepatic stage. | In pre-anhepatic stage, an average of 4 hours.
  Clot Formation Time (CFT, in seconds), the time needed to increase clot firmness from 2 to 20 mm amplitude as detected by thromboelastometry during pre-anhepatic stage.
Clot Formation Time in anhepatic stage. | In anhepatic stage, an average of 2 hours.
  Clot Formation Time (CFT, in seconds), the time needed to increase clot firmness from 2 to 20 mm amplitude as detected by thromboelastometry during anhepatic stage.
Clot Formation Time after reperfusion. | After reperfusion, an average of 4 hours.
  Clot Formation Time (CFT, in seconds), the time needed to increase clot firmness from 2 to 20 mm amplitude as detected by thromboelastometry after reperfusion.
Clot Formation Time at the end of surgery | At the end of surgery, an average of 12 hours.
  Clot Formation Time (CFT, in seconds), the time needed to increase clot firmness from 2 to 20 mm amplitude as detected by thromboelastometry at the end of surgery.
Angle α preoperative. | Preoperative up to 1 day before surgery.
  Angle α, the angle of tangent at 2 mm amplitude (ANG α, in degrees) as detected by thromboelastometry preoperatively.
Angle α in pre-anhepatic stage. | In pre-anhepatic stage, an average of 4 hours.
  Angle α, the angle of tangent at 2 mm amplitude (ANG α, in degrees) as detected by thromboelastometry during pre-anhepatic stage.
Angle α in anhepatic stage. | In anhepatic stage, an average of 2 hours.
  Angle α, the angle of tangent at 2 mm amplitude (ANG α, in degrees) as detected by thromboelastometry during anhepatic stage.
Angle α after reperfusion. | After reperfusion, an average of 4 hours.
  Angle α, the angle of tangent at 2 mm amplitude (ANG α, in degrees) as detected by thromboelastometry after reperfusion.
Angle α at the end of surgery | At the end of surgery, an average of 12 hours.
  Angle α, the angle of tangent at 2 mm amplitude (ANG α, in degrees) as detected by thromboelastometry at the end of surgery.
Maximum Clot Firmness preoperative. | Preoperative up to 1 day before surgery.
  Maximum Clot Firmness (MCF, in millimeters), the maximum amplitude of clot firmness finally achieved as detected by thromboelastography preoperatively.
Maximum Clot Firmness in pre-anhepatic stage. | In pre-anhepatic stage, an average of 4 hours.
  Maximum Clot Firmness (MCF, in millimeters), the maximum amplitude of clot firmness finally achieved as detected by thromboelastography during pre-anhepatic stage.
Maximum Clot Firmness in anhepatic stage. | In anhepatic stage, an average of 2 hours.
  Maximum Clot Firmness (MCF, in millimeters), the maximum amplitude of clot firmness finally achieved as detected by thromboelastography during anhepatic stage.
Maximum Clot Firmness after reperfusion. | After reperfusion, an average of 4 hours.
  Maximum Clot Firmness (MCF, in millimeters), the maximum amplitude of clot firmness finally achieved as detected by thromboelastography after reperfusion.
Maximum Clot Firmness at the end of surgery. | At the end of surgery, an average of 12 hours.
  Maximum Clot Firmness (MCF, in millimeters), the maximum amplitude of clot firmness finally achieved as detected by thromboelastography at the end of surgery.
Warm ischemic time | during the surgery, an average of 2 hours
  in minutes
Length of ICU stay | after the surgery, an average of 1 month
  in days
Length of hospital stay | postoperative, an average of 1 month
  in days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed HH Amin, Principal Investigator — Assistant Lecturer; Fatma AA Ahmed, Study Chair — Professor; Eman AE Ahmed, Study Director — Assistant professor; Ghada MA Abdelhamid, Study Director — Lecturer
Locations (1):
- Assiut university, Asyut, Egypt